CLINICAL TRIAL: NCT03673579
Title: Clinical Evaluation of the "NICU Clinical Decision Support Dashboard"
Brief Title: Clinical Evaluation of the "NICU Clinical Decision Support Dashboard" - MHSB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business pivot caused termination of study before enrollment.
Sponsor: Philips Healthcare (Industry)
Collaborators: Memorial Hospital of South Bend (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PCMS-17-07-18.1-MHSB
Record Dates: First submitted 2018-09-10; First posted 2018-09-17 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Preterm Birth; Low; Birthweight, Extremely (999 Grams or Less); Neonatal Infection; Satisfaction; Stress; Chronic Lung Disease; Growth Acceleration; Adverse Event
Keywords: NICU; Developmental care; Neuroprotective; Technology
MeSH Terms: conditions — Premature Birth; Birth Weight; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Prospective control data will be collected before the study devices are installed in all the NICU rooms. At the point of clinical go-live, there will be a single intervention group that all parents/clinicians will have the opportunity to participate in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- NICU Dashboard: Parent (Experimental): The parental intervention group will have access to the parent application on the NICU Dashboard. Parents will be able to view basic information about their baby's condition, educational material, and track core measures and developmental milestones.
  Parents of NICU babies will be asked to complete questionnaires at baseline and within 48 hours of NICU discharge.
  Interventions: Device: NICU Dashboard
- Standard Care: Parent (No Intervention): The Parental Control group will receive standard of care without any study devices.
- NICU Dashboard: Clinician (Experimental): The Clinician group will have access to the NICU Dashboard, which presents information from the EHR, bedside monitoring, and other systems of record through a pre-released FDA Class 2 clinical decision support rule-based system, to assist the appropriate evidence-based guidelines be integrated with team workflows. Caregivers educate and coach parents to facilitate integrating them into their infant's care.
  NICU clinicians will be asked to complete questionnaires 1) prior to clinical go-live of the intervention (baseline), 2) at the study mid-way point, and 3) upon completion of parent recruitment.
  Interventions: Device: NICU Dashboard

INTERVENTIONS:
Device: NICU Dashboard — The NICU Dashboard is displayed on a touch screen display mounted to the wall or on a rolling cart that will be placed near the bedside. The Dashboard will integrate information from various hospital/device sources in order to provide clinicians with one location to access and collectively interpret clinical findings and environmental factors. Parents will have their own view on the Dashboard that will allow them view their baby's progress, view educational materials, and have access to other resources at their fingertips.
  Other Names: Lotus Dashboard
  Arms: NICU Dashboard: Clinician; NICU Dashboard: Parent

SUMMARY:
This study evaluates the use of a NICU clinical integration system (Dashboard and accessories) in improving the quality of care delivered, patient health outcomes, and parent and clinician satisfaction. Clinicians will be asked to follow their current standard of care practices with the aid of this technology. About half of participants will receive care in NICU rooms with the Dashboard installed while the other half will receive standard care without the Dashboard.

DETAILED DESCRIPTION:
The current NICU environment can be stressful and overwhelming for parents of babies admitted and for clinicians caring for the babies. There is a wide range of monitors in a very clinical environment that does not take into account the comfort of neonates.

The Dashboard works in parallel with EHR and systems of record, and provides a cohesive view of the patient's status and planned clinical workflow in a single location for both parents and staff. Accessories such as environmental sensors and cameras are used to ensure that the environment is comfortable and promotes optimal development of the baby. Caregivers can educate and coach parents to facilitate integrating them into their infant's care. The NICU Dashboard also supports a family view to facilitate education and assist the family in tracking core measures and developmental milestones.

ELIGIBILITY:
NEONATES AND THEIR PARENTS

Inclusion Criteria:

* Admission to the NICU
* At least one parent (biological, guardian, or adoptive) involved
* One parent can understand and speak the English language
* Parent aged 18 years or older
* Parent with sufficient mental capacity to provide written informed consent as determined by a RN
* Signed informed consent from the parent

Exclusion Criteria:

* Expected discharge from the NICU in <48 hours

CLINICIANS INTERACTING WITH THE NICU DASHBOARD

Inclusion Criteria:

* Employee of institution with direct patient care in the NICU (e.g. physician, NP, RN, therapist)
* Expected interaction with the NICU Dashboard
* Signed informed consent

Exclusion Criteria:

* No interaction with the NICU Dashboard

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Rate of neonatal adverse events | Through study completion, an average of 1 year
  Preventable adverse events (e.g. unplanned extubations, medication errors)

SECONDARY OUTCOMES:
Incidence rate of Chronic Lung Disease | Through study completion, an average of 1 year
  Diagnosis
Rate of Readmission | 7 days and 30 days post-hospital discharge
  Number of readmissions (within 7 and 30 days) to a hospital over the number of total babies
Baby growth velocity | From date of NICU admission until the date of NICU discharge, assessed daily up to 365 days
  Rate of weight gain
Percent of time noise levels are within range | From date of NICU admission until the date of NICU discharge, assessed daily up to 365 days
  Hours that noise levels are within range over total patient-time
NICU Length of Stay | From date of NICU admission until the date of NICU discharge, assessed up to 365 days
  Days spent in the NICU from admission to discharge
Baby to parent skin-to-skin time | From date of NICU admission until the date of NICU discharge, assessed daily up to 365 days
  Self-reported time parents are performing skin-to-skin (kangaroo care), averaged
Parental Stressor Scale:NICU (PSS:NICU) | Upon signing informed consent (baseline) and within 96 hours of discharge
  For NICU parents 26-item questionnaire broken down into three constructs (Parental Role Alterations, Sights and Sounds of the Unit, and Infant Behavior and Appearance) designed to measure parental perception of stressors arising from the physical and psychosocial environment of the neonatal intensive care unit.
  1. = Not at all stressful (the experience did not cause you to feel upset, tense, or anxious)
  2. = A little stressful
  3. = Moderately stressful
  4. = Very stressful
  5. = Extremely stressful Total score will be calculated by summing each item score and averaged for the group. Each subscale will also be computed by summing the items within the subscale and averaging for each group.
  Higher scores represent worse outcomes
Neonatal Index of Parent Satisfaction (NIPS) | Within 96 hours of discharge
  For NICU parents 30-item questionnaire measuring parents' satisfaction with the care their newborn child receives while in a neonatal intensive care unit (NICU).
  7-point Likert-scale (1) lowest satisfaction to (7) highest satisfaction. Sum item scores to calculate total score, with lower scores corresponding to worse outcomes.
System Usability Scale (SUS) | Six months after study initiation (mid-point) and 12 months after study initiation (completion)
  For NICU parents and clinicians 10-item questionnaire with 2 constructs: usability and learnability 5-point Likert-scale (1) strongly disagree to (5) strongly agree The participant's scores for each question added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking. Based on research, a SUS score above a 68 would be considered above average and anything below 68 is below average, however the best way to interpret your results involves "normalizing" the scores to produce a percentile ranking.
The Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) Survey | Within 96 hours of discharge
  For NICU parents 7-item questionnaire assessing communication with doctors (4-items) and nurses (3-items).
  4-point Likert-scale: Never, Sometimes, Usually, Always The number of "Always" ratings for each participant is summed then divided by the number of items. The mean is then taken, stratified by group.
  Higher scores represent better outcomes.
Emotional Exhaustion Scale | Baseline (before study initiation), six months after study initiation (mid-point) and 12 months after study initiation (completion)
  For Clinicians only 4-item questionnaire about job-related frustrations. 4-point Likert-scale: (1) Disagree strongly to (5) Agree strongly. Item scores are summed and averaged by group. Higher scores represent worse outcomes.
Teamwork Perceptions Questionnaire (T-TPQ) | Baseline (before study initiation), six months after study initiation (mid-point) and 12 months after study initiation (completion)
  For Clinicians only 21-item questionnaire measuring 3 constructs: team function, mutual support, and communication 5 - Strongly Agree 4 - Agree 3 - Neutral 2 - Disagree
  1 - Strongly A total score is calculated for each teamwork construct. Summing scores in this manner allows for more accurate statistical testing.
  High scores indicate better outcomes.
Frequency of Missed Care (MISSCARE) | Baseline (before study initiation), six months after study initiation (mid-point) and 12 months after study initiation (completion)
  For Clinicians only 35-item questionnaire assessing the frequency that elements of nursing care are missed by nursing staff on the unit.
  1. - Always missed
  2. - Frequently missed
  3. - Occasionally missed
  4. - Rarely missed
  5. - Never missed Scores will be averaged per item, and a total MISSCARE score will be computed per individual by averaging all items.
  Higher scores represent better outcomes.
NASA Task Load Index (NASA-TLX) | Baseline (before study initiation), six months after study initiation (mid-point) and 12 months after study initiation (completion)
  For Clinicians only 6-item survey that rates perceived workload in order to assess the current workload in the NICU.
  Increments of high, medium and low estimates for each point results in 21 gradations on the scales assessing mental demand, physical demand, temporal demand, performance, effort, and frustration.
  Averages for each subscale will be computed. Higher scores represent worse outcomes.
Percent of time light levels are within range | From date of NICU admission until the date of NICU discharge, assessed daily up to 365 days
  Hours that light (lux) levels are within range over total patient-time

OTHER OUTCOMES:
Incidence of Hospital Acquired Infections | From date of NICU admission until the date of NICU discharge, assessed up to 365 days
  For example, CLABSI, Sepsis, VAP
Hand washing compliance rate | One year prior to study initiation, and through study completion, an average of one year
  Number of events found during audits
Cost of care | One year prior to study initiation, and through study completion, an average of one year
  Hospitalization costs (paid by insurance), costs/# of labs ordered, costs/# of images ordered

CONTACTS AND LOCATIONS:
Overall Officials: Robert White, MD, Principal Investigator — Memorial Hospital of South Bend, Mednax
Locations (1):
- Memorial Hospital of South Bend, South Bend, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
At this moment, Philips has no intention to share IPD with other researchers except those from institutions participating in this clinical investigation.